CLINICAL TRIAL: NCT06768138
Title: Intra-Arterial Thrombolysis After SUCCESSful Angiographic Recanalization in Acute Large Vessel Occlusion Stroke of the Anterior Circulation: the IA-SUCCESS Multicenter, Randomized Clinical Trial
Brief Title: Intra-Arterial Thrombolysis After SUCCESSful Reperfusion in Anterior Circulation Ischemic Stroke
Acronym: IA-SUCCESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Benjamin GORY, MD, PhD, Principal Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020PI054; 2023-506935-14-01 (EU CTIS Number)
Record Dates: First submitted 2024-12-13; First posted 2025-01-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Acute Ischemic
Keywords: Ischemic stroke; Thrombectomy; Endovascular treatment; Intra-arterial thrombolysis; Randomized controlled trial; Recanalisation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint will be assessed by central, independent blinded and qualified nurse certified in the assessment of the modified Rankin Scale (mRS) following a structured questionnaire of the mRS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunct intra-arterial thrombolysis (Experimental): Adjunct intra-arterial thrombolysis with Alteplase 0.225mg/kg after intravenous thrombolysis intravenous thrombolysis alone, bridging therapy, or mechanical thrombectomy alone.
  Interventions: Drug: Intra-arterial infusion of Alteplase
- No intra-arterial thrombolysis (No Intervention): Control group: no intra-arterial thrombolysis after intravenous thrombolysis alone, bridging therapy, or mechanical thrombectomy alone (according to standard of care).

INTERVENTIONS:
Drug: Intra-arterial infusion of Alteplase — Patients enrolled in the experimental arm will receive intra-arterial thrombolysis with Alteplase. The dose of Intra-arterial Alteplase is 0.225 mg/kg body weight with a maximal dose of 20 mg
  Arms: Adjunct intra-arterial thrombolysis

SUMMARY:
Stroke is a leading cause of disability and mortality worldwide. Despite the clinical benefit of mechanical thrombectomy, 1 out of 2 patients treated are functionally independent at 90 days. Achieving the best possible angiographic reperfusion is a key determinant of clinical outcome in acute ischemic stroke patients with anterior circulation large vessel occlusion. Mechanical thrombectomy is standard treatment for large vessel occlusion stroke patients within 24. In the setting of successful (eTICI ≥2b), adjunct intra-arterial thrombolysis may be a promising therapeutic option allowing recanalization of distal arterial occlusions (not accessible to mechanical devices) and improvement of upstream brain reperfusion by targeting microvascular obstruction.

The IA-SUCCESS randomized trial aims to assess the clinical and safety of adjunct intra-arterial thrombolysis vs. no adjunct intra-arterial thrombolysis after successful angiographic reperfusion in patients with acute anterior circulation large vessel occlusion stroke.

DETAILED DESCRIPTION:
Prospective phase 3 multicenter with open label blinded endpoint (PROBE) superiority randomized controlled trial, with health-economics evaluation.

The study strategy is to demonstrate the superiority of adjunct intra-arterial thrombolysis compared to no adjunct intra-arterial thrombolysis after successful angiographic reperfusion (eTICI 2b-2c-3) after intravenous alone, bridging therapy, or mechanical thrombectomy alone on 90-day functional outcome rate (shift of 90-day modified Rankin Scale toward a better functional outcome).

Patients with anterior circulation large vessel occlusion stroke will be recruited in the angiosuite by neurologists and/or neuroradiologists in participating centres after acute reperfusion therapy (intravenous thrombolysis alone, bridging therapy, or mecanical thrombectomy alone).

Patients enrolled in the experimental arm will receive intra-arterial thrombolysis with Alteplase. The dose of intra-arterial Alteplase is 0.225 mg/kg body weight and the maximal allowed dose is 20mg. Intra-arterial Alteplase will be injected through the guiding catheter placed in the internal carotid artery during 15 minutes.The total intra-arterial dose must be injected in the absence of complications.

Secondary objectives:

1. To assess the clinical and safety of adjunct intra-arterial thrombolysis.
2. To assess the cost-effectiveness of adjunct intra-arterial thrombolysis.
3. To assess the budget impact of new stroke management strategy in case of successful angiographic reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pre-stroke mRS 0-2
* Acute ischemic stroke with anterior circulation large vessel occlusion defined as intracranial internal carotid artery, M1, or M2 occlusion proven on CT or MRI
* NIHSS score ≥ 5 at admission
* Acute reperfusion strategy started within 24h after stroke onset according to the international guidelines
* DWI-ASPECTS ≥ 2 (MRI) or CT-ASPECTS ≥ 3
* Delay from imaging to puncture within 3 hours for transferred patients
* eTICI 2b-2c-3 after intravenous thrombolysis alone, bridging therapy, or mechanical thrombectomy alone and confirmed by catheter angiogram
* Person affiliated to or beneficiary of a social security plan

Exclusion Criteria:

* Person who do not speak French
* Contraindications for intra-arterial thrombolysis: Platelet count <100 000/mm3, INR >1.7, AOD use <48h or biological confirmation of activity and effective heparin treatment
* Bleeding-risk complications during the mechanical thrombectomy procedure (e.g carotid dissection, complicated femoral approach)
* Bleeding-risk complications consecutive to a fall associated with stroke
* More than 5 thrombectomy device
* Intracerebral hemorrhage
* Occlusion or high grade stenosis treated by stenting
* Patient expected to be unable to present or be available for 3-month visit follow-up
* Participation in another clinical trial within 30 days prior to the inclusion which the experiment may affect the 90-day mRS score
* Woman of childbearing age without effective contraception
* Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-09-16 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
The superiority of adjunct intra-arterial thrombolysis versus no adjunct intra-arterial thrombolysis | 90 (±15) days
  The primary endpoint is the severity of disability according to the distribution of scores on the modified Rankin Scale (mRS): mRS 0 to 6

SECONDARY OUTCOMES:
To assess the efficacy of adjunct intra-arterial thrombolysis | 90 (±15) days
  Distribution of the mRS score (0 to 6)
To assess the efficacy of adjunct intra-arterial thrombolysis | 90 (±15) days
  Excellent functional outcome (mRS 0-1)
To assess the efficacy of adjunct intra-arterial thrombolysis | 24 (±6) hours
  Early neurological improvement (reduction in National Institutes of Health Stroke Scale (NIHSS) score by at least 8 points, or NIHSS score of 0-1)
To assess the safety of adjunct intra-arterial thrombolysis | 24 (±6) hours
  Symptomatic and asymptomatic intracerebral hemorrhage within 24-hour on imaging follow-up, according to the Heidelberg classification (imaging core laboratory).
To assess the cost-effectiveness of adjunct intra-arterial thrombolysis | 12 months
  Incremental cost-effectiveness and cost-utility ratios of a strategy based on adjunct intra-arterial thrombolysis in case of successful angiographic reperfusion.
To assess the budget impact of new stroke management strategy in case of successful angiographic reperfusion | 12 months
  Total cost of each treatment strategy and net impact on the National Health Insurance System (difference in costs).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France